CLINICAL TRIAL: NCT03210714
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) - Phase 2 Subprotocol of Erdafitinib in Patients With Tumors Harboring FGFR1/2/3/4 Alterations
Brief Title: Erdafitinib in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With FGFR Mutations (A Pediatric MATCH Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01159; NCI-2017-01159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621B (Other: Children's Oncology Group); APEC1621B (Other: CTEP); U10CA180886 (NIH); UM1CA081457 (NIH)
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm; Recurrent Childhood Ependymoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Medulloblastoma; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Childhood Osteosarcoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Hepatoblastoma; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Glioma; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Recurrent Primary Central Nervous System Neoplasm; Recurrent Rhabdoid Tumor; Refractory Childhood Malignant Germ Cell Tumor; Refractory Childhood Osteosarcoma; Refractory Childhood Rhabdomyosarcoma; Refractory Childhood Soft Tissue Sarcoma; Refractory Ependymoma; Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Refractory Hepatoblastoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Glioma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Central Nervous System Neoplasm; Refractory Rhabdoid Tumor; Wilms Tumor
MeSH Terms: conditions — Familial ependymoma; Medulloblastoma; Neuroectodermal Tumors, Primitive, Peripheral; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Glioma; Neuroblastoma; Central Nervous System Neoplasms; Rhabdoid Tumor; Ependymoma; Lymphoma, Non-Hodgkin; Wilms Tumor | interventions — Specimen Handling; Biopsy; erdafitinib; Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (erdafitinib) (Experimental): Patients receive erdafitinib PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, PET scan, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Erdafitinib; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Procedure: Radionuclide Imaging; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo a bone marrow aspiration and/or biopsy
Procedure: Bone Scan — Undergo a bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ 42756493; JNJ-42756493; JNJ42756493
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Radionuclide Imaging — Undergo radionuclide imaging
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II Pediatric MATCH trial studies how well erdafitinib works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with FGFR mutations that have spread to other places in the body and have come back or do not respond to treatment. Erdafitinib may stop the growth of cancer cells with FGFR mutations by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with erdafitinib with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor genetic alterations in the FGFR1/2/3/4 pathway.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with erdafitinib with advanced solid tumors (including CNS tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor genetic alterations in the FGFR1/2/3/4.

II. To obtain information about the tolerability of erdafitinib in children with relapsed or refractory cancer.

III. To provide preliminary estimates of the pharmacokinetics of erdafitinib in children with relapsed or refractory cancer.

EXPLORATORY OBJECTIVE:

I. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive erdafitinib orally (PO) once daily (QD) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI), positron emission tomography (PET) scan, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to molecular analysis for therapy choice (MATCH) to APEC1621B based on the presence of an actionable mutation as defined in APEC1621SC
* Patients must be >/= 12 months and =/< 21 years of age at the time of study enrollment
* Patients must have a body surface area >/= 0.53 m^2 at enrollment
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as lesion that is at minimum 10 mm in one dimension on standard MRI or CT

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >/= 50% for patients > 16 years of age and Lansky >/= 50 for patients =/< 16 years of age; Note: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; >/= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >/= 7 days after the last dose of agent
  * Antibodies: >/= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =/< 1
  * Corticosteroids: if used to modify immune adverse events related to prior therapy, >/= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >/= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >/= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >/= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >/= 42 days
  * Cellular therapy: >/= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * X-ray therapy (XRT)/external beam irradiation including protons: >/= 14 days after local XRT; >/= 150 days after TBI, craniospinal XRT or if radiation to >/= 50% of the pelvis; >/= 42 days if other substantial bone marrow (BM) radiation

    * Note: radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, iobenguane I-131 [131I-MIBG]): >/= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to erdafitinib or another FGFR inhibitor such as (but not limited to) AZD4547, BGJ398, BAY1163877, LY2874455
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >/= 1000/mm^3 (performed within 7 days prior to enrollment)
  * Platelet count >/= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (performed within 7 days prior to enrollment)
  * Hemoglobin >/= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions) (performed within 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive platelet or packed [p]RBC transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >/= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows (performed within 7 days prior to enrollment):

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): male 0.6; female 0.6
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): male 0.8; female 0.8
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): male 1; female 1
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): male 1.2; female 1.2
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): male 1.5; female 1.4
  * Age: >/= 16 years; maximum serum creatinine (mg/dL): male 1.7; female 1.4
* Bilirubin (sum of conjugated + unconjugated) =/< 1.5 x upper limit of normal (ULN) for age (performed within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =/< 135 U/L; (for the purpose of this study, the ULN for SGPT is 45 U/L) (performed within 7 days prior to enrollment)
* Serum albumin >/= 2 g/dL (performed within 7 days prior to enrollment)
* Corrected QT (QTc) interval =/< 480 milliseconds
* Pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest)
* Patients must be able to swallow intact tablets
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal studies; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method, while receiving study treatment and for 3 months after the last dose of erdafitinib; male subjects (with a partner of child-bearing potential) must use a condom with spermicide when sexually active and must not donate sperm from the first dose of study drug until 3 months after the last dose of study drug
* Concomitant medications

  * Corticosteroids: patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >/= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible
  * Anti-GVHD agents post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
  * CYP3A4 agents: patients who are currently receiving drugs that are strong inducers or inhibitors of CYP3A4 are not eligible; Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed
  * CYP2C9 agents: patients who are currently receiving drugs that are strong inducers or moderate inhibitors of CYP2C9 are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* A history of cardiovascular diseases: unstable angina, myocardial infarction, or known congestive heart failure class II-IV within the preceding 12 months; cerebrovascular accident or transient ischemic attack within the preceding 3 months, pulmonary embolism within the preceding 2 months
* A history of any of the following: sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes, cardiac arrest, Mobitz II second degree heart block or third degree heart block; known presence of dilated, hypertrophic, or restrictive cardiomyopathy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with significant ophthalmologic conditions (uncontrolled glaucoma, central serous retinopathy, history of retinal vein occlusion or retinal detachment, excluding patients with longstanding findings secondary to existing conditions) are not eligible, to be confirmed with baseline ophthalmologic exam; all patients must have a baseline ophthalmologic exam, including fundoscopy to confirm no significant ophthalmologic conditions are present

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Lee, Principal Investigator — Children's Oncology Group
Locations (116):
- United States (114):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Erdafitinib)
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 6
Not completed — Physician Decision | 1
Not completed — Progressive disease | 11
Not completed — Refusal by patient/parent/guardian | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Erdafitinib)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors).
Time Frame: Up to 2 years from study entry
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Erdafitinib)
Number analyzed (Participants) | 20
percentage of patients | 10 [3.3 to 26.2]

2. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or Higher Adverse Events
Description: Percentage of patients experiencing grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Time Frame: Up to 2 years from study entry
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the 6 month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Pharmacokinetic (PK) Parameters
Description: A descriptive analysis of PK parameters will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Time Frame: Pre-dose Cycle 2 Day 1; 1-hour post-dose Cycle 2 Day 1; 2-hour post dose Cycle 2, Day 1; 4-hour post-dose Cycle 2, Day 1; 6-8-hour post-dose, Cycle 2 Day 1; 24-hour post dose, Cycle 2, Day 2
Reporting Status: Not Posted, anticipated posting 2025-12

5. Other Pre Specified Outcome: Changes in Tumor Genomic Profile
Description: A descriptive analysis will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years from study entry.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (Erdafitinib)
All-Cause Mortality (participants affected / at risk) | 8/20
Serious Adverse Events (participants affected / at risk) | 10/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erdafitinib) (N=20)
Enterocolitis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Pain (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erdafitinib) (N=20)
Anemia (Blood and lymphatic system disorders) | 10
Sinus bradycardia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 3
Dry eye (Eye disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2
Generalized edema (General disorders) | 1
Hypothermia (General disorders) | 1
Pain (General disorders) | 3
Conjunctivitis (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Mucosal infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 10
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 11
Blood bicarbonate decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
GGT increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
Thyroid stimulating hormone increased (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Hypersomnia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Muscle weakness left-sided (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT03210714/Prot_SAP_000.pdf